CLINICAL TRIAL: NCT00987779
Title: An Open, Randomized, Crossover Study In Healthy Subjects To Assess The Bioequivalence Of Gabapentin Between Japanese Commercial Tablet And Japanese Commercial Image Liquid Formulation And The Effect Of Food On The Pharmacokinetics Of Japanese Commercial Image Liquid Formulation
Brief Title: Bioequivalence Study Of Gabapentin Between Tablet And Liquid Formulation And The Food Effect Study Of Liquid Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A9451168
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Bioequivalence study; Food effect study; Pharmacokinetics; Gabapentin
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period I: Tablet(400 mg single dose) (Experimental): Period I: Tablet in fasting state, Period II: Liquid formulation in fasting state, Period III: Liquid formulation in fed state
  Interventions: Drug: Gabapentin
- Period I: Liquid formulation(400 mg single dose) (Experimental): Period I: Liquid formulation in fasting state, Period II: Tablet in fasting state, Period III: Liquid formulation in fed state
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Period I: Tablet in fasting state(400 mg single dose on Day 1 only of each Period; subjects stay in clinic for a total of 4 days for each period), Period II: Liquid formulation in fasting state(400 mg single dose on Day 1 only of each Period; subjects stay in clinic for a total of 4 days for each period), Period III: Liquid formulation(400 mg single dose on Day 1 only of each Period; subjects stay in clinic for a total of 4 days for each period) in fed state
  Arms: Period I: Tablet(400 mg single dose)
Drug: Gabapentin — Period I: Liquid formulation in fasting state(400 mg single dose on Day 1 only of each Period; subjects stay in clinic for a total of 4 days for each period), Period II: Tablet in fasting state(400 mg single doseon Day 1 only of each Period; subjects stay in clinic for a total of 4 days for each period), Period III: Liquid formulation(400 mg single doseon Day 1 only of each Period; subjects stay in clinic for a total of 4 days for each period) in fed state
  Arms: Period I: Liquid formulation(400 mg single dose)

SUMMARY:
Primary objective for this study is to demonstrate bioequivalence between Japanese commercial tablet and Japanese commercial image liquid formulation. Secondary objective for this study is to estimate the food effect for Japanese commercial image liquid formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Endpoints - Primary: plasma Cmax and AUCt of gabapentin. - Secondary: plasma AUCinf, AUClast, Tmax, kel, MRT and t1/2 of gabapentin | dosing to 3 days

SECONDARY OUTCOMES:
Safety Endpoints - Adverse events and safety laboratory data | dosing to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451168&StudyName=Bioequivalence%20Study%20Of%20Gabapentin%20Between%20Tablet%20And%20Liquid%20Formulation%20And%20The%20Food%20Effect%20Study%20Of%20Liquid%20Formulation